CLINICAL TRIAL: NCT03315676
Title: RCT Using Bonopurazan or Esomeprazole in Patients With NSAIDs-induced Erosions and/or Ulcers
Brief Title: Efficacy of Proton Pump Inhibitors in Gastrointestinal Erosions and/or Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Lecturer at Shinshu University School of Medicine, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPI 2017
Record Dates: First submitted 2017-10-07; First posted 2017-10-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Erosions and/or Ulcers
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Bonoprazan (Active Comparator): Daily intake of Bonoprazan
  Interventions: Drug: Oral Bonoprazan
- Oral Esomeprazol (Active Comparator): Daily intake of Esomeprazol
  Interventions: Drug: Oral Esomeprazol

INTERVENTIONS:
Drug: Oral Bonoprazan — To examine the efficacy of oral Bonoprazan in patients with NSAIDs-induced Erosions and/or Ulcers
  Arms: Oral Bonoprazan
Drug: Oral Esomeprazol — To examine the efficacy of oral Esomeprazol in patients with NSAIDs-induced Erosions and/or Ulcers
  Arms: Oral Esomeprazol

SUMMARY:
The aim of this study is to collect the data of clinical efficacy and safety after the usage of bonoprazon and esomeprazole when the patients take NSAIDs more than 2 weeks and have gastrointestinal symptoms who have had gastrointestinal erosions and/or ulcers in the past.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NSAIDs-induced gastrointestinal Erosions and/or Ulcers who want to take Bonoprazan or Esomeprazole

Exclusion Criteria:

* Patients allergic to Bonoprazan or Esomeprazole

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients are separately analyzed
Enrollment: 124 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-11-21 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with healing of gastrointestinal erosions and/or ulcers using major forceps | Change from Baseline Gastrointestinal erosions and/or ulcers at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan